CLINICAL TRIAL: NCT01398085
Title: Is Ablative Radio-iodine Necessary for Low Risk Differentiated Thyroid Cancer Patients
Brief Title: IoN- Is Ablative Radio-iodine Necessary for Low Risk Differentiated Thyroid Cancer Patients
Acronym: IoN
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/10/0299; 2011-000144-21 (EudraCT Number); Cancer Research UK (Other Grant/Funding Number: CRUK/11/010); ISRCTN (Registry Identifier: ISRCTN80416929)
Record Dates: First submitted 2011-07-06; First posted 2011-07-20 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Thyroid Cancer
Keywords: Papillary thyroid carcinoma; Follicular thyroid carcinoma; Hurthle cell carcinoma of the thyroid; Iodine Radioisotopes
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary; Adenocarcinoma, Follicular; Thyroid cancer, Hurthle cell | interventions — Sodium Iodide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radioactive iodine (RAI) ablation Arm (Active Comparator): Patients will be randomised to receive Radioactive iodine (RAI) ablation I131 1.1 GBq
  Interventions: Radiation: I131 1.1 GBq
- No Radioactive iodine (No-RAI) ablation (No Intervention): Patients will be randomised to receive No Radioactive iodine (No-RAI) ablation

INTERVENTIONS:
Radiation: I131 1.1 GBq — Radio-iodine
  Other Names: Sodium iodide capsule
  Arms: Radioactive iodine (RAI) ablation Arm

SUMMARY:
IoN is a phase II/ III trial that will look to ascertain whether or not radio-iodine ablation is necessary for low risk differentiated thyroid cancer patients.

DETAILED DESCRIPTION:
Phase II: to determine if recruitment into a phase III trial is feasible, with a target of 10 patients per month during a minimum of 6 months (evaluated within months 7-18 of the trial).

Phase III: to determine whether the 5-year disease-free survival rate among patients who do not have routine Radioactive iodine (RAI) ablation is non-inferior to those who do.

ELIGIBILITY:
TNM eligibility is assessed against TNM7 (7th edition 2009) or TNM8 (8th edition 2017, in use in the UK from 01/01/2018).

Eligibility Criteria using TNM7:

Inclusion criteria:

* Histological confirmation of well differentiated thyroid carcinoma: MDT decision for inclusion based on overall clinico-pathological assessment is critical.
* R0 total thyroidectomy (in one or two stages, no residual disease present; Rx at the discretion of the MDT) within the last 6 months
* Negative pregnancy test in women of child bearing potential
* Aged 16 or over
* WHO performance status 0 - 2, self-caring
* Histological confirmation of differentiated thyroid carcinoma:MDT decision for inclusion based on overall clinico-pathological assessment
* Papillary thyroid cancer (PTC):

  * Non aggressive histological features (small foci of aggressive histology allowed at the discretion of the MDT)
  * pT1a (≤1cm) unifocal with positive level VI lymph nodes (pN1a)
  * pT1a(m): all individual foci ≤1cm
  * pT1b and pT1b(m): >1-2cm
  * pT2 and pT2(m): >2-4cm
  * pT3 and pT3(m): >4cm confined to the thyroid
  * pT3 R0 +/- (m): any size with minimal ETE if recommended by the MDT
  * pN0
  * pN1a
  * pNX
* Follicular thyroid cancer (FTC) (including oncocytic or Hürthle cell cancer):

  o minimally invasive FTC -which are considered low risk and are recommended by the specialist MDT based on overall clinico-pathological assessment
  * pT1b and pT2: >1-4cm intrathyroidal
  * pT3 R0:any size up to 4 cm with minimal ETE if recommended by the MDT
* Histological material available for Central Review (see section 9.7)
* Willing to use contraception for the duration of the trial until 6 months post radioiodine treatment (for females) or 4 months post treatment (for males) (see section 6.4.2), if allocated to the ablation group.

NB: Multifocal tumours (≥2 foci) of all histological types should be designated with "(m)", and the size of the largest focus determines the classification (as described in the TNM 7th edition). For example, if there are two foci, one 0.8cm and the other 3cm, the classification is based on the 3cm focus; i.e. pT2(m).

Exclusion criteria:

* pT1a - Papillary and Follicular carcinoma which is unifocal and ≤1cm in size, without any positive nodes or unfavourable clinical features, treated by lobectomy.
* Up to 4cm non-invasive Encapsulated Follicular Variant of Papillary Thyroid Cancer (eFVPTC) with no capsular or vascular invasion (>4 cm can be included at the discretion of the MDT)
* non-invasive follicular tumour with papillary-like nuclei (NIFTP)
* Anaplastic, poorly differentiated or medullary carcinoma
* R1 or R2 thyroidectomy
* Patients with:

  * pN1b
  * M1
* Aggressive Papillary thyroid cancer with any of the following features:

  * Widely invasive
  * Poorly differentiated
  * Anaplastic
  * Tall cell
  * Columnar cell
  * Diffuse sclerosing variants
* Follicular thyroid cancer/Hürthle cell cancer with any of the following features:

  * Tumours greater than 4cm
  * Widely invasive
  * Poorly differentiated
  * Anaplastic
* Incomplete resection or lobectomy
* pT4a and pT4b or macroscopic and microscopic tumour invasion of loco-regional tissues or structures
* Pregnant women or women who are breast feeding
* Patients who have had CT performed with iv contrast less than 2-3 months before ablation
* Previous treatment for thyroid cancer (except surgery in last 6 months)
* Previous malignancies with limited life expectancy or likely to interfere with the patient's ability to be able to comply with treatment and/or follow-up for at least 5 years
* The following GI conditions: dysphagia, oesophageal stricture, active gastritis, gastric erosions, peptic ulcer, suspected reduced gastrointestinal motility
* MDT decision against ablation or suitability for trial in light of severe co-morbid condition/s including:

  * Unstable angina
  * Recent myocardial infarction or cerebrovascular accident (CVA)
  * Severe labile hypertension
  * Any patient who cannot comply with radiation protection including:

    * patients with learning difficulties
    * patients with dementia
    * patients with a tracheostomy that require nursing care
    * patients requiring frequent nursing/ medical supervision

Eligibility Criteria using TNM8:

Inclusion criteria:

* Histological confirmation of well differentiated thyroid carcinoma: MDT decision for inclusion based on overall clinico-pathological assessment is critical.
* R0 total thyroidectomy (in one or two stages, no residual disease present; Rx at the discretion of the MDT) within the last 6 months
* Negative pregnancy test in women of child bearing potential
* Aged 16 or over
* WHO performance status 0 - 2, self-caring
* Histological confirmation of differentiated thyroid carcinoma:MDT decision for inclusion based on overall clinico-pathological assessment
* Papillary thyroid cancer (PTC):

  * Non aggressive histological features (small foci of aggressive histology allowed at the discretion of the MDT)
  * pT1a (≤1cm) unifocal with positive level VI lymph nodes (pN1a)
  * pT1a(m): all individual foci ≤1cm
  * pT1b and pT1b(m): >1-2cm
  * pT2 and pT2(m): >2-4cm
  * pT3a and pT3a(m): >4cm confined to thyroid
  * pT1a/1b/2/3 (where minimal microscopic extra thyroidal extension (ETE) does not change the T score) +/- (m): any size with minimal ETE if recommended by the MDT
  * pN0
  * pN1a
  * pNX
* Follicular thyroid cancer (FTC) (including oncocytic or Hürthle cell cancer):

  o minimally invasive FTC -which are considered low risk and are recommended by the specialist MDT based on overall clinico-pathological assessment
  * pT1b and pT2: >1-4cm intrathyroidal
  * pT1a/1b/2/3a (where minimal microscopic ETE does not change the T score): any size up to 4 cm with minimal ETE if recommended by the MDT
* Histological material available for Central Review (see section 9.7)
* Willing to use contraception for the duration of the trial until 6 months post radioiodine treatment (for females) or 4 months post treatment (for males) (see section 6.4.2), if allocated to the ablation group.

Exclusion criteria:

* pT1a - Papillary and Follicular carcinoma which is unifocal and ≤1cm in size, without any positive nodes or unfavourable clinical features, treated by lobectomy.
* Up to 4cm non-invasive Encapsulated Follicular Variant of Papillary Thyroid Cancer (eFVPTC) with no capsular or vascular invasion (>4 cm can be included at the discretion of the MDT)
* non-invasive follicular tumour with papillary-like nuclei (NIFTP)
* Anaplastic, poorly differentiated or medullary carcinoma
* R1 or R2 thyroidectomy
* Patients with:

  * pN1a with level VII involvement
  * pN1b
  * M1
* Aggressive Papillary thyroid cancer with any of the following features:

  * Widely invasive
  * Poorly differentiated
  * Anaplastic
  * Tall cell
  * Columnar cell
  * Diffuse sclerosing variants
* Follicular thyroid cancer/Hürthle cell cancer with any of the following features:

  * Tumours greater than 4cm
  * Widely invasive
  * Poorly differentiated
  * Anaplastic
* Incomplete resection or lobectomy
* pT3b, pT4a and pT4b or macroscopic and microscopic tumour invasion of loco-regional tissues or structures
* Pregnant women or women who are breast feeding
* Patients who have had CT performed with iv contrast less than 2-3 months before ablation
* Previous treatment for thyroid cancer (except surgery in last 6 months)
* Previous malignancies with limited life expectancy or likely to interfere with the patient's ability to be able to comply with treatment and/or follow-up for at least 5 years
* The following GI conditions: dysphagia, oesophageal stricture, active gastritis, gastric erosions, peptic ulcer, suspected reduced gastrointestinal motility
* MDT decision against ablation or suitability for trial in light of severe co-morbid condition/s including:

  * Unstable angina
  * Recent myocardial infarction or cerebrovascular accident (CVA)
  * Severe labile hypertension
  * Any patient who cannot comply with radiation protection including:

    * patients with learning difficulties
    * patients with dementia
    * patients with a tracheostomy that require nursing care
    * patients requiring frequent nursing/ medical supervision

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2012-05; Primary Completion 2024-12 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Phase II: monthly patient accrual rates | Evaluated within months 7-18 of the trial
  To determine if recruitment into a phase III trial is feasible
Phase III: Disease-free thyroid specific survival | From randomisation until recurrence or death from thyroid cancer
  DFS measured from randomisation until date of recurrence or death from thyroid cancer

SECONDARY OUTCOMES:
Phase III: Mortality (cause and date of death) | From randomisation until death
  Cause and date of death
Phase III: Occurrence of loco-regional recurrence or metastatic disease | After follow up is complete (estimated year 8-9 of trial)
  Both groups will be compared to ascertain if radio-iodine results in a statistically significant reduction in risk in developing loco-regional recurrence in the low risk subgroup of patients.
Phase III: Stage of cancer at the time of recurrence, and the ability to treat this successfully | After follow up is complete (estimated year 8-9 of trial)
  Both groups will be compared to ascertain if radio-iodine results in a statistically significant difference in the stage of cancer at the time of recurrence, and the ability to treat this successfully.
Phase III: Health-related quality of life | After follow up is complete (estimated year 8-9 of trial)
  Quality of Life
Phase III: Adverse events for all patients | After follow up is complete (estimated year 8-9 of trial)
  Adverse events will be collected for patients in both groups during treatment and the groups compared during analysis.
Phase III: Further neck surgery | After follow up is complete (estimated year 8-9 of trial)
  The number of further neck surgeries will be collected for patients in both groups during follow up and the groups compared during analysis.
Phase III: Further RAI ablations | After follow up is complete (estimated year 8-9 of trial)
  Further RAI ablation and the reasons for this
Phase III: Cost-effectiveness | After follow up is complete (estimated year 8-9 of trial)
  Costs of treatment for both groups will be collected for duration of trial to see if there is a difference between the two.

CONTACTS AND LOCATIONS:
Overall Officials: Ujjal Mallick, MBBS, Master of Surgery, FRCR, Principal Investigator — Newcastle-upon-Tyne Hospitals NHS Foundation Trust
Locations (32):
- United Kingdom (32):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - University Hospital Bristol NHS Foundation Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - East Kent Hospitals University NHS Foundation Trust, Canterbury
  - Mid Essex Hospitals Services NHS Trust, Chelmsford
  - Gloucestershire Hospitals NHS Trust, Cheltenham
  - Royal Derby hospital NHS foundation trust, Derby
  - NHS Lothian, Edinburgh
  - Royal Devon and Exeter NHS Trust, Exeter
  - Glasgow and Clyde NHS Trust, Glasgow
  - The Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - Ipswich Hospital NHS Trust, Ipswich
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - Royal Marsden NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Barts Health NHS Trust, London
  - Guys and St Thomas' NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Maidstone and Tunbridge Wells NHS Trust, Maidstone
  - The Christie NHS Foundation Trust, Manchester
  - South Tees Hospitals NHS Trust, Middlesbrough
  - Velindre NHS Trust, Nantgarw
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Norfolk and Norwich University Hospitals NHS Trust, Norwich
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Southend University Hospitals NHS Trust, Southend
  - East and North Herts, Stevenage
  - Royal Wolverhampton NHS Trust, Wolverhampton

REFERENCES:
- [Derived] Mallick U, Newbold K, Beasley M, Garcez K, Wadsley J, Johnson SJ, Stephenson T, Gaze M, Goodman A, Jefferies S, Sivabalasingham S, Slevin N, Wilkinson DP, Macias-Fernandez E, Power D, Roques T, Speed L, Nutting C, Mochloulis G, Gerrard G, Candish C, Morgan S, Tripathi D, Truran P, Arthur C, Wieczorek A, Madhavan K, Maclean J, Boote D, Kim D, Pascoe A, Pitiyage G, Forsyth S, Ambrose E, Chang E, Farnell K, Hackshaw A. Thyroidectomy with or without postoperative radioiodine for patients with low-risk differentiated thyroid cancer in the UK (IoN): a randomised, multicentre, non-inferiority trial. Lancet. 2025 Jul 5;406(10498):52-62. doi: 10.1016/S0140-6736(25)00629-4. Epub 2025 Jun 18. PMID 40543520
- See also: Cancer Research UK & UCL Cancer Trials Centre website — http://www.ctc.ucl.ac.uk/